CLINICAL TRIAL: NCT04044898
Title: A Pharmacokinetics and Safety Study of Aminolevulinic Acid Hydrochloride Topical Powder in Subjects With Moderate to Severe Facial Acne Vulgaris.
Brief Title: Pharmacokinetics and Safety of ALA in Acne Vulgaris
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Shanghai Fudan-Zhangjiang Bio-Pharmaceutical Co., Ltd. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: F0014-ALA-201811
Record Dates: First submitted 2019-08-01; First posted 2019-08-05 (Actual); Last update posted 2022-03-17 (Actual); Status verified 2022-03

CONDITIONS: Acne Vulgaris
Keywords: Acne vulgaris
MeSH Terms: conditions — Acne Vulgaris

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Low dose (Experimental)
  Interventions: Drug: ALA 5%
- High dose (Experimental)
  Interventions: Drug: ALA 10%

INTERVENTIONS:
Drug: ALA 5% — prepare 5% ALA solution, apply topically to the affected area for 1.5 hours, single dose
  Arms: Low dose
Drug: ALA 10% — prepare 10% ALA solution, apply topically to the affected area for 3 hours, single dose
  Arms: High dose

SUMMARY:
This study will evaluate the pharmacokinetics and safety of ALA in patients with moderate and severe acne vulgaris after single dose in different dosages.

ELIGIBILITY:
Inclusion Criteria:

1. Male and female subjects between 18 and 45 years of age (all subjects are male in pilot study);
2. Diagnosis of moderate to severe facial acne vulgaris by the clinician according to the Pillsbury International Improvement Classification III-IV criteria;
3. Body weight≥50 kg, body mass index (BMI) ≥19 and ≤28 kg/m2；
4. Subjects (including male subjects) voluntarily adopt effective physical contraception from 14 days prior to the use of the study drug to 1 month after the end of the study, and have no fertility or donation of sperm/egg plan;
5. Subjects voluntarily sign informed consent forms after being informed of the study procedures，requirements and possible adverse reactions of the study drug.

Exclusion Criteria:

1. Suffer from allergic diseases ，suspect or known to have porphyrin disease or known to be allergic to test medication and/or porphyrin， or allergic persons (such as allergies to two or more drugs, food or pollen);
2. Allergies to visible light
3. Secondary acne patients, such as acne caused by occupational acne and corticosteroids.
4. Suffering from malignant tumors and suffering from diseases such as heart, endocrine, blood, liver, immunity, metabolism, urinary system, lungs, nervous system, rheumatism/joint, mental, kidney, etc led the researchers to believe that the subject is not suitable for participating in this study
5. Have been treated with systemic Vitamin A acid drugs therapy within 2 months before the study and/or antibiotics or hormonal drugs within 4 weeks before the study
6. Used local topical vitamin A acid drugs within the 4 weeks before the study or patients with topical antibiotics, glucocorticoid and other topical treatment of acne drugs within the 2 weeks before the study
7. Vaccination within 4 weeks prior to the use of the study drug;
8. Severe external injuries were suffered within the first 3 months (90 days) prior to the use of the study drug, or Patients who have undergone surgical treatment may significantly affect the process of studying drugs in vivo or safety assessment;
9. Taked clinical trial drugs within 3 months (90 days) prior to the use of the study drug, or be participating in or plan to participate in other clinical trials during the study period.
10. Drinking alcohol regularly within 3 months (90 days) prior to the use of the study drug (≥3 times a week, and the average drink is equivalent to 50° white wine ≥200 mL) or can not quit drinking during the study, or alcohol breath test positive
11. Smoking cigarettes (more than 10 cigarettes or equivalent of tobacco per day) within 3 months (90 days) prior to the use of the study drug or those who cannot quit smoking during the study;
12. Blood loss/blood donation more than 300 mL (except for female physiological blood loss), blood transfusion or blood product use within 3 months (90 days) prior to the use of the study drug, or plan to be blood donors during the study period or 1 month after the end of the study l (30 days) )
13. Consumed excessively daily tea, coffee or caffeinated beverages (up to 8 cups per day, 200 mL per cup) within 1 month (30 days) prior to the use of the study drug;
14. Drinks or food intake excessive of alcohol or caffeine (coffee, tea, cola, chocolate, etc.) within 48 hours prior to the use of the study drug ;
15. Have a history of drug abuse or positive drug abuse screening;
16. Hepatitis B surface antigen or hepatitis C virus antibody or treponema pallidum antibody positive or HIV Screening positive;
17. Physical examination (except acne), Vital Signs, laboratory examination (blood routine, urine routine, liver function, renal function, fasting blood glucose, blood lipids, etc).and 12 lead ECG results were judged to be abnormal and clinically significant by clinicians
18. Pregnant or lactating female; blood or urine pregnancy test positive
19. Have a history of blood or Needles fainting, or difficulty in collecting blood
20. Unable to complete the study for other reasons or Researchers believe that those who should not be included;
21. Researchers and their relatives including spouses and children will be not allowed to participate in this study.

Ages: 18 Years to 45 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 19 (Actual)
Dates: Start 2021-01-12 (Actual); Primary Completion 2021-07-30 (Actual); Study Completion 2021-12-06 (Actual)

PRIMARY OUTCOMES:
Maximum Plasma Concentration [Cmax] | 24 hours postdose
  pharmacokinetic parameter
Area Under the Curve [AUC] | 24 hours postdose
  pharmacokinetic parameter
Tmax | 24 hours postdose
  pharmacokinetic parameter
Half-life Time [T1/2] | 24 hours postdose
  pharmacokinetic parameter
Clearance [CL] | 24 hours postdose
  pharmacokinetic parameter
Apparent Volume of Distribution [Vd] | 24 hours postdose
  pharmacokinetic parameter
Maximum Plasma Concentration [Cmax](after deduction of background) | 24 hours postdose
  pharmacokinetic parameter
Area Under the Curve [AUC](after deduction of background) | 24 hours postdose
  pharmacokinetic parameter
Tmax(after deduction of background) | 24 hours postdose
  pharmacokinetic parameter
Half-life Time [T1/2](after deduction of background) | 24 hours postdose
  pharmacokinetic parameter
Clearance [CL](after deduction of background) | 24 hours postdose
  pharmacokinetic parameter
Apparent Volume of Distribution [Vd](after deduction of background) | 24 hours postdose
  pharmacokinetic parameter
Incidence of adverse events | 2 days postdose
  Number of participants with treatment related adverse events as assessed by physical examination, vital signs, clinical laboratory values, local skin responses

CONTACTS AND LOCATIONS:
Locations (1):
- Huashan Hospital, Shanghai, Shanghai Municipality, China

IPD SHARING:
Plan to Share IPD: No